CLINICAL TRIAL: NCT06870266
Title: Comparison of Pregnancy Rates in Modified Natural Frozen Embryo Transfer (FET) Cycle After Luteal Support with GnRH Agonist Versus Progesterone: Prospective Randomized Study
Brief Title: Comparison of Pregnancy Rates in Modified Natural Frozen Embryo Transfer (FET) Cycle After Luteal Support with GnRH Agonist Versus Progesterone
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Yael Lerner, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0357-24-SZMC
Record Dates: First submitted 2025-02-20; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Ivf; Frozen Embryo Transfer (FET)
MeSH Terms: conditions — Long Qt Syndrome 3 | interventions — Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SYNAREL (Active Comparator): LUTEAL PHASE SUPPORT WITH SYNAREL 200 MCG X2 DAY
  Interventions: Drug: Nafarelin nasal spray
- UTEROGESTAN (Active Comparator): LUTEAL PHASE SUPPORT WITH UTEROGESTAN 200 MG X2 DAY
  Interventions: Drug: Utrogestan®

INTERVENTIONS:
Drug: Nafarelin nasal spray — NAFARLIN 200 MCG X2 DAY
  Arms: SYNAREL
Drug: Utrogestan® — UTROGESTAN 200 MG X2 DAY
  Arms: UTEROGESTAN

SUMMARY:
Background:

The capability to transfer frozen embryos reduces embryo loss following in vitro fertilization (IVF) and results in higher pregnancy rates compared to a single IVF cycle.

Endogenous progesterone from the corpus luteum, following frozen embryo transfer in natural or modified natural cycles, is expected to provide sufficient luteal support, as observed in spontaneous pregnancies. Nevertheless, research has demonstrated higher pregnancy success rates with additional luteal support. The current standard for luteal phase support involves vaginal progesterone administration.

Several case reports have indicated that administering a gonadotropin-releasing hormone (GnRH) agonist during the luteal phase does not compromise pregnancy continuation achieved through IVF and may, in fact, enhance implantation success.

Studies have shown that the luteal phase can be maintained with a GnRH agonist alone, without the need for progesterone supplementation.

A recent prospective randomized controlled trial compared standard progesterone support with GnRH agonist support in fresh embryo transfers. The group receiving GnRH agonist support demonstrated a significantly higher pregnancy rate.

Given the studies proving the positive impact of GnRH agonist, there is a need for a prospective randomized controlled trial to evaluate the use of GnRH agonist support in frozen embryo transfers.

Aims and Significance:

This study aims to compare pregnancy rates between women receiving GnRH agonist treatment and those receiving standard progesterone-based luteal support during frozen embryo transfers in natural cycles as part of IVF treatments.

Conducting a prospective comparative study will enable us to assess the effectiveness of GnRH agonist treatment relative to standard luteal phase support. Based on the results, the investigators may consider treatment with intranasal GnRH agonist, which improves quality of life and may also enhance pregnancy and live birth rates.

Methods:

The study will be conducted on patients scheduled to undergo modified natural cycles. Participants will be randomly allocated into two groups:

1. Study Group: Luteal phase support will begin on the day of ovulation with Nafarelin nasal spray (200 mcg twice daily) for two weeks, until pregnancy blood test (hCG).
2. Control Group: Luteal phase support will be provided through vaginal progesterone. Endometrin 100 mg twice daily. If the hCG test is positive, the supportive treatment will continue until the 8th week of pregnancy, as per the attending physician's instructions.

Clinical follow-up will include monitoring for clinical pregnancy outcomes, miscarriage rates, and live births.

DETAILED DESCRIPTION:
Background:

The ability to transfer frozen embryos allows for the storage of embryos created during in vitro fertilization (IVF) treatments for later use. Frozen embryo transfers offer several advantages, such as reducing embryo loss following IVF and achieving higher pregnancy rates compared to a single IVF cycle. The rate of frozen embryo transfers has increased in recent years due to the growing trend of single embryo transfer (SET) in young women, the use of preimplantation genetic testing (PGT), and the prevention of ovarian hyperstimulation syndrome (OHSS). With recent advances in cryopreservation technology, embryo freezing offers the aforementioned benefits without compromising pregnancy rates.

There are several methods for preparing the endometrium for frozen embryo transfer:

1. Natural Cycle (NC) - Timing ovulation by detecting the LH surge. The advantage of the natural cycle is the body's natural preparation for implantation without the need for medical intervention. However, its disadvantages include the need for close monitoring to detect ovulation and the inflexibility of embryo transfer timing, leading to a higher rate of cycle cancellations.
2. Modified Natural Cycle (mNC) - Inducing ovulation using an hCG trigger injection. This method provides slightly greater flexibility in scheduling the embryo transfer according to clinical availability, reducing patient visits and improving convenience.
3. Medicated Cycle - Preparing the endometrium with exogenous estrogen and progesterone. This method is suitable for women with irregular ovulation, offering greater flexibility and fewer cycle cancellations.

Studies comparing natural and modified natural cycles have yielded inconclusive results.

Endogenous progesterone from the corpus luteum after natural ovulation is expected to provide adequate luteal support, similar to that in spontaneous pregnancies. Therefore, theoretically, luteal support may not be necessary in frozen embryo transfers during natural cycles. However, the benefit of luteal support remains controversial.

A meta-analysis published in Human Reproduction in 2021 evaluated the effect of progesterone luteal support, showing higher pregnancy rates in the group that received support compared to those that did not. It is noteworthy that most studies involved ovulation induced by hCG (mNC).

Several case reports from the 1990s demonstrated that the unintentional administration of GnRH agonists during the luteal phase did not impair ongoing pregnancies achieved through IVF and might even support implantation. The mechanism by which GnRH agonists improve implantation rates remains unclear. Proposed mechanisms include luteal support by stimulating LH secretion from gonadotrophic cells in the pituitary gland, direct effects on the endometrium and embryo through GnRH receptors, and regulation of hCG production and secretion by the preimplantation placenta and embryo.

Indeed, a systematic review by Cochrane published in 2015 showed that adding GnRH agonists to progesterone luteal support increased pregnancy and live birth rates.

In 2006, Pirrard hypothesized that the luteal phase could be maintained with GnRH agonists alone, without the need for progesterone. After feasibility and pilot studies published in 2005 and 2006, a randomized controlled trial (RCT) was conducted in 2015 comparing the effectiveness of GnRH agonist-only luteal support with standard vaginal progesterone therapy. Although the sample size was small, the study reported higher implantation and pregnancy rates in the GnRH agonist group, but statistical significance was not reached.

In 2017, a retrospective study was published comparing 1,093 cycles with GnRH agonist support to 1,436 cycles with standard progesterone support. The study aimed to assess live birth rates while improving patient quality of life during treatment. The GnRH agonist group showed higher mid-luteal progesterone levels and significantly higher live birth rates. Although the groups were not comparable, as the GnRH agonist group included younger women and those undergoing fewer cycles, the higher live birth rate remained statistically significant even after adjusting for age, treatment cycle, BMI, and obstetric history.

It is important to note that GnRH agonists are not considered teratogenic. In over 340 women exposed to GnRH agonists during the mid-luteal phase, the rates of congenital anomalies (2.5%) and miscarriage (15%) were similar to the general IVF population.

A prospective randomized controlled trial conducted at Shaare Zedek Medical Center and published in 2023 compared standard progesterone support to GnRH agonist support in fresh embryo transfers. The study included 127 cycles evenly divided between the two groups. The group receiving GnRH agonist support demonstrated a significantly higher pregnancy rate.

Given the studies demonstrating the positive impact of GnRH agonist on pregnancy and live birth rates in fresh embryo transfers, there is a need for a prospective randomized controlled trial evaluating GnRH agonist support in frozen embryo transfers.

Aims & Significance:

The aim of this study is to compare pregnancy rates between women treated with a GnRH agonist and those receiving standard progesterone-based luteal support in frozen embryo transfers during natural cycles as part of IVF treatments.

Primary Outcome:

• Clinical pregnancy rate (presence of an embryo with a heartbeat on ultrasound)

Secondary Outcomes:

• Positive pregnancy test rate (hCG), implantation rate (gestational sac), live birth rate, early miscarriage, and late miscarriage Conducting a prospective comparative study will enable an assessment of the efficacy of GnRH agonist-only treatment relative to standard luteal phase support. Based on the findings, intranasal GnRH agonist may be considered as a therapeutic option that improves patient quality of life and potentially enhances pregnancy and live birth rates.

Research Plan:

During the dedicated clinic visit for frozen embryo transfer cycles, demographic and clinical data will be collected. Women meeting the inclusion criteria (undergoing a modified natural cycle) will receive an explanation of the study's purpose and sign an informed consent form in accordance with institutional Helsinki Committee regulations.

The number of embryos to be transferred will be determined based on the woman's age. Participants will be randomly assigned to one of the two study groups using a computer-generated 1:1 randomization process. Sealed envelopes containing information about the assigned luteal support protocol will be attached to the consent forms, ensuring allocation concealment.

Participants will be monitored in the IVF unit with blood tests and ultrasound scans to identify the dominant follicle. Once the follicle reaches a diameter of at least 17 mm, a single dose of hCG (Ovitrelle 250 mcg) will be administered to induce ovulation.

Embryo Transfer: The timing of the transfer will depend on the age of the frozen embryo. For a 3-day-old embryo, transfer will occur 5 days after the hCG injection.

Study Group:

Treatment will begin 48 hours after the hCG injection (Day 0) with Nafarelin nasal spray (200 mcg twice daily) for two weeks following ovulation induction, up to the pregnancy blood test (hCG).

Control Group:

Luteal support will be provided with vaginal progesterone, either Endometrin 100 mg twice daily or Utrogestan 200 mg twice daily. If the hCG test is positive, supportive treatment will continue until the 8th week of pregnancy, according to the attending physician's instructions.

Clinical pregnancy will be defined as the presence of an embryo with a heartbeat on ultrasound. Pregnancy outcomes will be determined through a phone consultation with the patient 9 months after the treatment. Pregnancy termination will be classified as early or late miscarriage or live birth.

Setting:

The study will be conducted in the IVF Unit of the Department of Obstetrics and Gynecology at Shaare Zedek Medical Center.

Sample Size:

A total of 150 patients will be randomly allocated into two groups.

Inclusion Criteria:

1. Women treated at the Shaare Zedek IVF clinic scheduled for frozen embryo transfer
2. Normo-ovulatory women
3. Women undergoing frozen embryo transfer in a modified natural cycle
4. Age 18-40
5. BMI 18-35

Exclusion Criteria:

1. Women undergoing medicated FET cycles
2. BMI >35 or <18
3. Women with hydrosalpinx
4. Women with congenital or acquired uterine anomalies (e.g., myomas)
5. Egg donation or surrogacy
6. Women with endometriosis
7. Intolerance to GnRH agonists
8. Nasal congestion or respiratory conditions affecting nasal absorption

Statistical Methods:

Based on the clinical pregnancy rates observed in the previous RCT conducted in our department, a sample size of 127 participants was sufficient to demonstrate a statistically significant difference in clinical pregnancy rates between the two luteal support methods. Therefore, it was decided to recruit approximately 150 patients for this study.

Categorical variables will be compared using the Chi-square test, while continuous variables will be compared using Student's t-test or Mann-Whitney U test, depending on the distribution (normal vs. non-normal). A multivariate regression analysis will be performed to identify independent factors associated with clinical outcomes. Statistical significance will be defined as a p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Women treated at the Shaare Zedek IVF clinic scheduled for frozen embryo transfer
2. Normo-ovulatory women
3. Women undergoing frozen embryo transfer in a modified natural cycle
4. BMI 18-35
5. Age 18-40

Exclusion Criteria:

1. Women undergoing medicated FET cycles
2. BMI >35 or <18
3. Women with hydrosalpinx
4. Women with congenital or acquired uterine anomalies (e.g., myomas)
5. Egg donation or surrogacy
6. Women with endometriosis
7. Intolerance to GnRH agonists
8. Nasal congestion or respiratory conditions affecting nasal absorption

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | two months after ET
  positive fetal heart beat

SECONDARY OUTCOMES:
positive pregancny | two weeks after ET
  positive hcg levels (>25 IU\L)
implantation rate | two months after ET
  eveidence of gestational sac in the uterus
live birth rate | 9 months after the treatment
  live birth after 24 weeks pregnancy
miscarriage rate | up to 24 weeks pregnancy
  miscarriage before 24 weeks pregnancy

IPD SHARING:
Plan to Share IPD: No